CLINICAL TRIAL: NCT06151106
Title: A Multicenter, Prospective and Single-arm Clinical Study on the Treatment of Refractory/Relapsed Peripheral T-cell Lymphoma (R/R PTCL) With Chidamide and Duvalisib
Brief Title: Chidamide and Duvalisibon for the Treatment of Refractory/Relapsed Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Dongguan People's Hospital (Other Government); Huizhou Municipal Central Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Sun Yat-sen University (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-02
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Peripheral T Cell Lymphoma; Relapsed Peripheral T-Cell Lymphoma; Refractory T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined with Duvillisib (Experimental)
  Interventions: Drug: Chidamide combined with Duvillisib

INTERVENTIONS:
Drug: Chidamide combined with Duvillisib — Specified dose on specified days

SUMMARY:
To determine the efficacy and safety of Chidamide combined with Duvalisib in the treatment of refractory/relapsed peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
This is a Phase 2, open-label clinical trial study that aims to evaluate the efficacy (Overall Response Rate, Complete Response, Partial Response, Overall Survival, Progression Free Survival) and adverse effects of Chidamide combined with Duvalisib in the treatment of refractory/relapsed peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Peripheral T-cell lymphoma (PTCL) or NK/T-cell lymphoma confirmed by histopathology/cytology according to the classification standard of the World Health Organization in 2008
2. Relapsed and refractory patients who have received at least first-line systemic treatment with anthracycline-containing drugs in the past. Recurrence is defined as relapse after CR or progression after PR, SD. The refractory disease was defined as previous systemic chemotherapy, PD in response evaluation for 2 cycles or SD in response evaluation for 4 cycles.
3. There must be at least one evaluable or measurable lesion meeting Lugano2014 standard: lymph node lesion and the measurable lymph node length should be > 1.5cm;
4. Patients aged at 18-75 years old;
5. ECOG 0-2
6. Routine blood examination: absolute neutrophil count ≥ 1.5× 10 9/L, platelet ≥ 75x10 9/L, Hb ≥ 80g/L.
7. Expected survival ≥3 months 8 No radiotherapy, chemotherapy, targeted therapy, or hematopoietic stem cell transplantation was received within 4 weeks before enrollment.

9. The patient or his/her legal representative must provide written informed consent before carrying out any special inspection or procedure of the study.

Exclusion Criteria:

1. Patients with central nervous system (CNS) or meningeal invasion
2. Any of the following laboratory abnormalities: absolute neutrophil count (ANC) < 1.5× 10*9/L, Hb< 80 g/L, PLT < 75×10 9 /L, organ dysfunction, are defined as follows: total bilirubin (TBiL) > 1.5 upper limit of normal value (ULN), or AST or ALT >2.5ULN, except the following situations. if patients with liver infiltrated by lymphoma cells, AST and ALT < 5ULN could be enrolled.
3. International normalized ratio (INR)>1.5ULN or partially activated prothrombin time (APTT) > 1.5 ULN
4. The active infection of human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) should be excluded except for the following patients: patients with HBV infection (HBsAg or HBcAg positive) but HBV DNA negative. These patients need continuous antiviral treatment and HBV DNA PCR detection every cycle. additionally, patients with HCV serology positive but HCV RNA negative can be enrolled.
5. In patients with CMV infection (IgM positive), CMV DNA was positive by PCR.
6. Meet any of the following criteria related to visceral function: all kinds of clinically significant abnormal rhythm or conduction need clinical pre-diagnosis Hereditary QT interval syndrome or QTcF>480 msec or taking drugs that may cause Qt interval delay or torsade de pointes. A variety of clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina, and coronary artery bypass grafting in the first 6 months of the group, with New York's cardiology (NYHA) classification of grade 3 or above. Left ventricular ejection fraction (LVEF )<40%, or uncontrolled blood pressure controlled by drugs (Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mgHg).
7. Have a history of stroke or intracranial hemorrhage within 6 months before drug administration for the first time
8. Major surgery was performed within 4 weeks before drug administration for the first study
9. Any PI3K inhibitor has been used before and the disease has progressed during the treatment period (within 6 months after the last use)
10. Received systemic anti-tumor therapy or radiotherapy within 4 weeks before the first study drug administration
11. The last time you participated in clinical trials of other drugs before the administration of the first study drug was less than 2 weeks or the last time you used targeted drugs (such as antibody drugs) was less than 4 weeks
12. patients received the transplantation of somatic hematopoietic stem cells within 3 months before the first drug administration
13. Patients received allogeneic hematopoietic stem cell transplantation or having any active graft-versus-host disease within 6 months before first drug administration.
14. Take a strong inducer or inhibitor of cytochrome P4503A4 (CYP3A4) within 2 weeks before drug administration (3 weeks for Hypericum perforatum) for the first time.
15. Before the first enrollment, the toxic reaction of previous anti-tumor therapy has not recovered to ≤1 level (except alopecia).
16. Patients with uncontrolled systemic infection requiring intravenous antibiotic treatment
17. Currently suffering from other primary tumors that need active treatment according to the guidelines
18. Inability to take drugs orally, previous surgical history or serious gastrointestinal diseases such as dysphagia and active gastric ulcer may affect the absorption of drugs
19. Pregnant (serum pregnancy test results are positive) or lactating women
20. Any other diseases, abnormal metabolism, abnormal physical examination or abnormal laboratory examination with significant clinical significance, according to the researcher's judgment, it is reasonable to suspect that the patient has a certain disease or state that is not suitable for using these two drugs, or it will affect the interpretation of the research results or put the patient in a high-risk situation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 27 months
  Percentage of participants with best overall response of partial response (PR) and complete response (CR), using the Lugano criteria.
Complete Response Rate | Up to 27 months
  Complete response (CR) is evaluated according to the Lugano criteria for lymphoma response.

SECONDARY OUTCOMES:
Partial Response Rate | Up to 27 months
  Partial response (PR) is evaluated according to the Lugano criteria for lymphoma response.
Progression Free Survival | Up to 27 months
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall Survival | Up to 27 months
  OS will be measured from the date of registration to the date of the event (i.e., death) or the date of last follow-up to evaluate that event. Patients who are event-free at their last follow-up evaluation will be censored at that time point.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- The First Affiliated Hosptial of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No